CLINICAL TRIAL: NCT00713700
Title: Closure of Patent Ductus Arteriosus With the AMPLATZER DUCT Occluder II
Brief Title: AMPLATZER Duct Occluder II Clinical Study
Acronym: ADO II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL00233
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Patent Ductus Arteriosus
Keywords: patent ductus arteriosus; PDA
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device (Experimental)
  Interventions: Device: AMPLATZER Duct Occluder II

INTERVENTIONS:
Device: AMPLATZER Duct Occluder II — AMPLATZER Duct Occluder II

SUMMARY:
The objective of this study is to investigate the safety and effectiveness of the ADO II in patients with a PDA.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have diagnosis of a PDA
* Subject must have a PDA < 5.5mm in diameter by angiography
* Subject must have a PDA < 12mm in length by angiography
* Subject must have a PDA > 3mm in length by angiography
* Subject/legally authorized representative must give consent to participate in the clinical study
* Subject/legally authorized representative must consent to follow-up for the duration of the clinical study

Exclusion Criteria:

* Subject must not be < 6 kilograms for the procedure
* Subject must not be < 6 months of age
* Subject must not be ≥ 18 years of age
* Subject must not have a descending aorta < 10mm in diameter
* Subject must not have a right to left shunt through the patent ductus arteriosus
* Subject must not have PVR above 8 Woods units or a Rp/Rs >0.4
* Subject must not have intracardiac thrombus
* Subject must not have additional cardiac anomalies requiring surgical or interventional correction
* Subject must not have history of more than two lower respiratory infections within the last year (i.e., pneumonia)
* Subject must not have active infection requiring treatment at the time of implant
* Subject must not have contraindication to anticoagulation treatment
* Female subjects of child bearing age must not be pregnant or desire to become pregnant within six months post implant*
* Subject must not be participating in another study for an investigational drug and/or device that may clinically interfere with this study's endpoints

  * If the subject desires to become pregnant after six months post-implant, further restriction is at the discretion of their physician.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Actual)
Dates: Start 2008-08; Primary Completion 2011-10 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Children's Hospital and Health Center, San Diego, California
  - University of California San Francisco Hospital, San Francisco, California
  - The Children's Hospital - Denver, Aurora, Colorado
  - Alfred I. DuPont Hospital for Children -Nemours Cardiac Center, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Memorial Regional Hospital (Joe DiMaggio Children's Hospital), Hollywood, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - The Children's Hospital Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital at Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas SW Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Device: AMPLATZER Duct Occluder II : AMPLATZER Duct Occluder II
Period: Overall Study
Arm/Group | Device
Started | 192
Completed | 188
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Device
Number analyzed (Participants) | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 192
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 72
Region of Enrollment [Number; unit: participants]
  United States | 192

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint is the Rate of Device and Procedure Related Serious Adverse Events (SAE) 180 Days Post Procedure.
Description: The primary safety endpoint is the rate of device and/or procedure related SAEs reported in subjects whom device placement is attempted from the procedure through 180 days post procedure
  SAEs are defined as: Adverse events resulting in the following; death, life-threatening adverse event, inpatient hospitalization or prolongation of existing hospital stay, persistent or significant disability/incapacity or medically significant event.
Time Frame: 180 days
Population: Of the 192 enrolled subjects, 188 completed follow-up through 180 days post procedure;3 subjects were lost to follow-up (LTFU) before the 180-day interval and 1 subject was discontinued at the end of the 6-month visit without follow-up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Device
Number analyzed (Participants) | 188
percentage of participants | 1.6 [.33 to 4.59]

2. Primary Outcome: The Primary Effectiveness Endpoint is the Rate of Complete Closure of the Ductus Arteriosus at the Six-month Follow-up.
Description: The primary efficacy endpoint is the rate of complete closure of the ductus arteriosus as assessed by the absence of residual flow and continuous murmur at the six-month follow-up by transthoracic echocardiography and physical exam respectively.
Time Frame: 180 days
Population: Of the 192 enrolled, 178 subjects experienced successful device placement.Of the 178 subjects with the device implanted,166 had a 6-month TTE and physical examination before 200 days post procedure or had an explant before the 6-month follow-up interval ended.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Device
Number analyzed (Participants) | 166
percentage of participants | 98.19 [94.81 to 99.63]

ADVERSE EVENTS:
Arm/Group | Device
Serious Adverse Events (participants affected / at risk) | 3/192
Other Adverse Events (participants affected / at risk) | 19/192
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=192)
Device Embolization (Injury, poisoning and procedural complications) | 1 (1)
Residual shunt requiring closure (Surgical and medical procedures) | 2 (2)
Sinus tachycardia (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Device (N=192)
Pain (General disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other